CLINICAL TRIAL: NCT05988554
Title: Efficacy Testing of Hibiscus Sabdariffa Extract and Collagen Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 23-048-B
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Skin Condition
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo sachet (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo sachet
- Hibiscus sabdariffa extract and collagen products (Experimental)
  Interventions: Dietary Supplement: Hibiscus sabdariffa extract and collagen products

INTERVENTIONS:
Dietary Supplement: Placebo sachet — Consume 1 sachet daily
  Arms: Placebo sachet
Dietary Supplement: Hibiscus sabdariffa extract and collagen products — Consume 1 sachet daily
  Other Names: SPRING Collagen Powder
  Arms: Hibiscus sabdariffa extract and collagen products

SUMMARY:
To assess Hibiscus sabdariffa extract and collagen products on skin condition improvement

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged above 20 years old

Exclusion Criteria:

* Subject who is not willing to participate in this study.
* Patients with diseases of the skin, liver, kidney.
* Subjects who have known cosmetic, drug or food allergies, difficulty in digestive tract absorption or disorder.
* Female who is pregnant or nursing or planning to become pregnant during the course of the study.
* Received facial laser therapy, chemical peeling or UV overexposure (> 3 hr/week) in the past 4 weeks.
* Constant drug use
* Students who are currently taking courses taught by the principal investigator of this trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
The change of skin collagen density | Week 0, week 4, week 8
  DermaLab® Series SkinLab Combo was utilized to measure skin pores. Units: arbitrary units
The change of skin wrinkles | Week 0, week 4, week 8
  VISIA Complexion Analysis System was utilized to measure skin wrinkles. Units: arbitrary units
The change of skin texture | Week 0, week 4, week 8
  VISIA Complexion Analysis System was utilized to measure skin texture. Units: arbitrary units
The change of skin elasticity | Week 0, week 4, week 8
  SoftPlus was utilized to measure skin elasticity. Units: arbitrary units
The change of skin moisture | Week 0, week 4, week 8
  Corneometer® CM825 was utilized to measure skin moisture. Units: arbitrary Corneometer® units 0-120

SECONDARY OUTCOMES:
The change of skin melanin index | Week 0, week 4, week 8
  Mexameter® MX18 was utilized to measure skin melanin index. Units: arbitrary units
The change of skin L* value | Week 0, week 4, week 8
  Chroma Meter MM500 was utilized to measure skin L* value. Units: arbitrary units, 0-100
The change of transepidermal water loss (TEWL) | Week 0, week 4, week 8
  Tewameter® TM 300 was utilized to measure TEWL. Units: g/hm²
The change of skin pores | Week 0, week 4, week 8
  VISIA Complexion Analysis System was utilized to measure skin pores. Units: arbitrary units
The change of skin spots | Week 0, week 4, week 8
  VISIA Complexion Analysis System was utilized to measure skin spots. Units: arbitrary units

OTHER OUTCOMES:
The change of self-assessment skin condition | Week 0, week 4, week 8
  A self-assessment questionnaire was collected to evaluate skin condition

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hua Liang, Principal Investigator — Chia Nan University of Pharmacy ＆ Science
Locations (1):
- Chia Nan University of Pharmacy ＆ Science, Tainan, Taiwan